CLINICAL TRIAL: NCT02574819
Title: Methylnaltrexone (MNTX) for Treatment of Opioid-induced Constipation in Advanced Illness Patients : a Multicenter, Randomized, Double-blind , Placebo-controlled Trail
Brief Title: Study of Methylnaltrexone in Opioid-Induced Constipation Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTTQ-MNTX
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Opioid-induced Constipation
Keywords: opioid-induced constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): Methylnaltrexone (MNTX) nearly 0.15mg/kg administered every other day for 2 weeks.
  Interventions: Drug: Methylnaltrexone (MNTX)
- Placebo (Placebo Comparator): Placebo administered every other day for 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone (MNTX) — MNTX nearly 0.15mg/kg administered every other day for 2 weeks. Baseline laxatives and rescue laxative ( enemas/suppositories ) were allowed, but could not be administered within 4 hours of the study drug.
  Arms: Drug
Drug: Placebo — Placebo administered every other day for 2 weeks. Baseline laxatives and rescue laxative ( enemas/suppositories ) were allowed, but could not be administered within 4 hours of the study drug.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind , placebo-controlled trail to investigate the safety and efficacy of subcutaneous methylnaltrexone for treating opioid-induced constipation in patients with advanced illness.

DETAILED DESCRIPTION:
Methylnaltrexone is a quaternary derivative of the pure opioid antagonists naltrexone. It is fairly lipid soluble and readily cross the blood-brain barrier. This property provides methylnaltrexone with the potential to block the undesired side-effects of opioid pain medications predominantly mediated by receptors located peripherally while sparing opioid effects mediated at receptors in the central nervous system, most importantly analgesia.

This is a multicenter, randomized, double-blind , placebo-controlled trail to investigate the safety and efficacy of subcutaneous methylnaltrexone for treating opioid-induced constipation in patients with advanced illness. The randomization schedule was used to assign patients in a 2:1 ratio to multicenter or an equal volume of placebo administered subcutaneously on alternate days for 2 weeks. The clinical trail was estimated to enroll 180 patients totally.

ELIGIBILITY:
Inclusion Criteria:

* A life expectancy of 3 month or more
* Qualifying patients received opioids for analgesia for 1 week or more and a stable regimen of opioids and laxatives for 3 or more days before study entry
* Patients had opioid-induced constipation with either fewer than three laxation during the preceding week and no clinically meaningful laxation (as determined by the in investigator ) within 24h before the first study dose or no clinically meaningful laxation within 48h before the first study dose
* During the two-week trail , patients would keep their life habits (dietary fiber , fluid intake and physical activity)
* Patients volunteered for the trail
* Women of childbearing potential had negative pregnancy tests. Both male and female patients need to take effective contraceptives to avoid pregnancy.

Exclusion Criteria:

* Constipation that was not primarily caused by opioids ( as determined by the investigator)
* Mechanical gastrointestinal obstruction, an indwelling peritoneal catheter, clinically active diverticular disease , fecal impaction , acute surgical abdomen , and fecal ostomy
* Patients had the surgery plan which would effect the results of pain assessment
* Patients had hypersensitivity to methylnaltrexone , naltrexone or naloxone or if any investigational drug or experimental product

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who had the Rescue-free laxation response within 4 hours of the initial dose | up to 4 hours
  Within 4 hours after the initial dose, if clinical significant bowel movement happened, the drug therapeutic effect was confirm. In the meantime, the time of bowel movement and other properties of bowel movement were recorded. The percentage of patients who had rescue-free laxation response is the primary outcome.

SECONDARY OUTCOMES:
The proportion of subjects who had at least 2 Rescue-free laxation responses within 4 hours after each doses from the first dose to the forth dose | up to 8 days
  Record the frequency of laxation. After 1-4 dose, within 4 hours of every dose, record the dose number when bowel movement happened
The proportion of subjects who had Rescue-free laxation response within 4 hours after each doses from the second dose to the last dose | up to 12 days
The proportion of subjects who had Rescue-free laxation response within 4-24h after each dose | up to 14 days
The proportion of subjects who had ≥3 laxation responses per week | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shiying Yu, Professor, Principal Investigator — Tongji Hospital in Wuhan
Locations (12):
- China (12):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Provincial cancer Hospital, Fuzhou, Fujian
  - Zhongnan Hospital of Wuhan University, Wuhan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Linyi Cancer Hospital, Linyi, Shandong
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xin Hua Hospital affiliated to Shanghai Jiao Tong University School of Medicine Chongming Branch, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xian, Shanxi
  - Tumor Hospital of Yunnan Province The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan